CLINICAL TRIAL: NCT06512129
Title: Phenotypes in Sepsis - Extracellular Water for Volume Status Characterization
Brief Title: Defining Volume Status in Sepsis With Extracellular Water Measurement
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-06866-01.1
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the influence of extracellular water on volume status in adult sepsis patients presenting with hemodynamic instability. The main question it aims to answer is:

• Can measurement of extracellular water (MoistureMeterD, Delfin Technologies Ltd, Kuopio, Finland) contribute to the description of hemodynamic instability in adult sepsis patients.

Patients with sepsis admitted to intensive care will receive standard care with the addition of measurement of extracellular water.

DETAILED DESCRIPTION:
Adult patients with sepsis admitted to any of our ICUs will be recruited. During the first three days after inclusion blood samples and extended non-invasive monitoring, including monitoring of the microcirculation (CytoCam) and measurement of extracellular water (dielectronic constant), will be added to routine care and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults with sepsis.

Exclusion Criteria:

* Pregnancy, other than sepsis known cause of shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to an ICU in Uppsala with suspected or confirmed sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Phenotypes in sepsis - extracellular water for volume status characterization. | 7 days
  Can measurement of extracellular water (MoistureMeterD, Delfin Technologies Ltd, Kuopio, Finland) contribute to the description of hemodynamic instability in adult sepsis patients during the first 72 hours?

CONTACTS AND LOCATIONS:
Overall Officials: Annelie Barrueta Tenhunen, MD, PhD, Principal Investigator — Uppsala University, Region Uppsala
Locations (1):
- AnOpIva, Uppsala, Uppsa, Sweden

IPD SHARING:
Plan to Share IPD: No
The data will only be accessible to the research team.

REFERENCES:
- [Background] Nuutinen J, Ikaheimo R, Lahtinen T. Validation of a new dielectric device to assess changes of tissue water in skin and subcutaneous fat. Physiol Meas. 2004 Apr;25(2):447-54. doi: 10.1088/0967-3334/25/2/004. PMID 15132310
- [Background] Toro C, Markarian B, Mayrovitz HN. Breast Cancer-Related Lymphedema Assessed via Tissue Dielectric Constant Measurements. Cureus. 2024 Apr 29;16(4):e59261. doi: 10.7759/cureus.59261. eCollection 2024 Apr. PMID 38813316
- [Background] De Backer D, Cecconi M, Chew MS, Hajjar L, Monnet X, Ospina-Tascon GA, Ostermann M, Pinsky MR, Vincent JL. A plea for personalization of the hemodynamic management of septic shock. Crit Care. 2022 Dec 1;26(1):372. doi: 10.1186/s13054-022-04255-y. PMID 36457089